CLINICAL TRIAL: NCT05787353
Title: Hospital- Versus Home-based Cardiopulmonary Rehabilitation for Post-acute COVID-19 Symptoms
Brief Title: Cardiopulmonary Rehabilitation for Post-acute COVID-19 Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir City Hospital (Other)
Responsible Party: Principal Investigator, Fulya Bakılan, Principal Investigator, Eskisehir City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CardioPulmonaryRehab
Record Dates: First submitted 2023-03-24; First posted 2023-03-28 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Cardiopulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home based cardiopulmonary rehabilitation group (Experimental): This was a retrospective study. 43 patients who had home based cardiopulmonary rehabilitation programme between January and July 2023, in our rehabilitation clinic.
  Interventions: Other: Exercise programme
- Hospital based cardiopulmonary rehabilitation group (Experimental): This was a retrospective study. 45 patients who had hospital based cardiopulmonary rehabilitation programme between January and July 2023, in our rehabilitation clinic.
  Interventions: Other: Exercise programme

INTERVENTIONS:
Other: Exercise programme — Both protocols consisted of aerobic, breathing and flexibility exercises. Hospital-based CPR: three or four days per week for a total of 20 sessions. Home-based CPR: three or four days/a week over a period of six weeks.

SUMMARY:
The purpose of this RETROSPECTIVE study was to compare the effect of a hospital and home-based cardiopulmonary rehabilitation (CPR) program on exercise endurance and quality of life in post-acute COVID-19 patients.

88 post-acute COVID-19 patients were divided two groups according to receiving hospital (n=45) or home-based CPR (n=43)in our rehabilitation clinic between January and July 2021. Both protocols consisted of aerobic, breathing and flexibility exercises. Hospital-based CPR: three or four days per week for a total of 20 sessions. Home-based CPR: three or four days/a week over a period of six weeks. The results of six meters walk test (6MWT) for exercise endurance as a main outcome measure, and Borg-dyspnea/fatigue, the visual analog scale (VAS) for pain and the Short Form-36 (SF-36) as secondary outcome measures before and after treatment were recorded.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older
* having COVID-19 treatment (home quarantine/hospital/intensive care unit) according to a positive polymerase chain reaction (PCR) test in a nasopharyngeal + oropharyngeal swab or chest computed tomography (CT)
* participating in a home-based exercise program (for 6 weeks) or hospital-based CPR (for 12-20 sessions) due to post-acute COVID-19 symptoms (fatigue, myalgia, dyspnea).

Exclusion Criteria:

* Patients who had both a negative PCR test and chest CT
* Patients who had not completed the six minute walk test (6MWT), Borg scales, Short Form-36 and Visual analog scale-pain.
* Acute COVID-19 patients (patients whose symptoms had started less than one month previous)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Exercise endurance | One day before exercise programme start and one day later exercise programme ends
  Six minutes walk test (All patients walked along a 30-meter-long corridor without obstacles at their normal walking speed, how many meters they walked was noted.)

SECONDARY OUTCOMES:
Dyspnea | One day before exercise programme start and one day later exercise programme ends
  Borg scale were also measured before and after 6MWT for perceived dyspnea (scale range from 0 to 10)
Muscle fatigue | One day before exercise programme start and one day later exercise programme ends
  Borg muscle fatigue (scale range from 6 to 20: higher values show more severe symptoms)
short form 36 | One day before exercise programme start and one day later exercise programme ends
  A quality-of-life assessment was performed using the Short Form-36, which has 36 items regarding physical function, physical role, emotional role, energy, body pain, mental health, general health, and social function. The scale ranges from 0 (poor health) to 100 (perfect health)
Musculoskeletal Pain | One day before exercise programme start and one day later exercise programme ends
  Visual analog scale-pain was used to measure general body musculoskeletal pain, which was assessed from 0 (no pain) to 10 (worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Fulya Bakılan, Assoc. Prof., Principal Investigator — Eskişehir Osmangazi University
Locations (1):
- Eskişehir Osmangazi University, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No